CLINICAL TRIAL: NCT02968771
Title: Metabolomic Profile of Patients Undergoing Myocardial Perfusion SPECT
Acronym: METS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: METS
Record Dates: First submitted 2016-11-16; First posted 2016-11-21 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Ischemic Heart Disease
Keywords: Coronary artery disease; Cardiac perfusion SPECT; Metabolomics
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples without DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with Physical Cardiac Stress: Patients with Physical Cardiac Stress
  Interventions: Other: Non intervention
- Patients with Physical and Pharmacological Cardiac Stress: Patients with Physical and Pharmacological Cardiac Stress with adenosine agonist
  Interventions: Other: Non intervention
- Patients with Pharmacological Cardiac Stress: Patients with Pharmacological Cardiac Stress with adenosine agonist
  Interventions: Other: Non intervention

INTERVENTIONS:
Other: Non intervention

SUMMARY:
The aim of this study is to analyze metabolomic pattern of patients after cardiac stress in order to detect differences based on the type of stress (physical or pharmacological with adenosine agonists) and result of test (positive or negative for ischemia) and to indentify biochemical markers with prognostic value. Clinical data of enrolled patients regarding demographics, cardiovascular risk factors, pretest probability and previous cardiovascular disease will be recorded. Follow up will be at one, three and five years and will be performed by clinical recordings or phone call when necessary. Blood samples of patients undergoing myocardial perfusion SPECT (Single Photon Emission Computed Tomography) are taken before, immediately after stress and 2h after stress. Serum samples will be analyzed by nuclear magnetic resonance in order to know metabolomic profile.

DETAILED DESCRIPTION:
The aim of this study is to analyze metabolomic pattern of patients after cardiac stress in order to detect differences based on the type of stress (physical or pharmacological with adenosine agonists) and result of test (positive or negative for ischemia) and to indentify biochemical markers with prognostic value. Clinical data of enrolled patients regarding demographics, cardiovascular risk factors, pretest probability and previous cardiovascular disease will be recorded. Follow up will be at one, three and five years and will be performed by clinical recordings or phone call when necessary. Blood samples of patients undergoing myocardial perfusion SPECT are taken before, immediately after stress and 2h after stress. Serum samples will be analyzed by nuclear magnetic resonance in order to know metabolomic profile.

ELIGIBILITY:
Inclusion Criteria:

* Patients men or women ≥ 18 years of age
* Patients with prescription of cardiac perfusion SPECT

Exclusion Criteria:

* Patients with loss of consciousness or confuse, not able to read the information and to sign the writting consent
* Pregnant women
* Patients with dobutamine indications in the stress protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prescription of cardiac perfusion SPECT
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Result of myocardial perfusion SPECT: positive or negative for angina, ischemia or perfusion defect. | 2 days
Metabolomic profile on NMR (Nuclear Magnetic Resonance ) analysis of serum sample | 6 month
  Once all samples analyzed, in order to identify of specific patterns associated to any group (type of test or result of test).

SECONDARY OUTCOMES:
Combined end point: Cardiovascular death, Myocardial infarction, Coronary revascularization. | 1 year
Combined end point: Cardiovascular death, Myocardial infarction, Coronary revascularization. | 3 years
Combined end point: Cardiovascular death, Myocardial infarction, Coronary revascularization. | 5 years
Angina treatment initiation | 1 year
Angina treatment initiation | 3 years
Angina treatment initiation | 5 years
Metabolomic profile on NMR analysis of serum sample | 1 year
Metabolomic profile on NMR analysis of serum sample | 3 years
Metabolomic profile on NMR analysis of serum sample | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Task Force Members; Montalescot G, Sechtem U, Achenbach S, Andreotti F, Arden C, Budaj A, Bugiardini R, Crea F, Cuisset T, Di Mario C, Ferreira JR, Gersh BJ, Gitt AK, Hulot JS, Marx N, Opie LH, Pfisterer M, Prescott E, Ruschitzka F, Sabate M, Senior R, Taggart DP, van der Wall EE, Vrints CJ; ESC Committee for Practice Guidelines; Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Knuuti J, Valgimigli M, Bueno H, Claeys MJ, Donner-Banzhoff N, Erol C, Frank H, Funck-Brentano C, Gaemperli O, Gonzalez-Juanatey JR, Hamilos M, Hasdai D, Husted S, James SK, Kervinen K, Kolh P, Kristensen SD, Lancellotti P, Maggioni AP, Piepoli MF, Pries AR, Romeo F, Ryden L, Simoons ML, Sirnes PA, Steg PG, Timmis A, Wijns W, Windecker S, Yildirir A, Zamorano JL. 2013 ESC guidelines on the management of stable coronary artery disease: the Task Force on the management of stable coronary artery disease of the European Society of Cardiology. Eur Heart J. 2013 Oct;34(38):2949-3003. doi: 10.1093/eurheartj/eht296. Epub 2013 Aug 30. No abstract available. PMID 23996286
- [Background] Liga R, Vontobel J, Rovai D, Marinelli M, Caselli C, Pietila M, Teresinska A, Aguade-Bruix S, Pizzi MN, Todiere G, Gimelli A, Chiappino D, Marraccini P, Schroeder S, Drosch T, Poddighe R, Casolo G, Anagnostopoulos C, Pugliese F, Rouzet F, Le Guludec D, Cappelli F, Valente S, Gensini GF, Zawaideh C, Capitanio S, Sambuceti G, Marsico F, Filardi PP, Fernandez-Golfin C, Rincon LM, Graner FP, de Graaf MA, Stehli J, Reyes E, Nkomo S, Maki M, Lorenzoni V, Turchetti G, Carpeggiani C, Puzzuoli S, Mangione M, Marcheschi P, Giannessi D, Nekolla S, Lombardi M, Sicari R, Scholte AJ, Zamorano JL, Underwood SR, Knuuti J, Kaufmann PA, Neglia D, Gaemperli O; EVINCI Study Investigators. Multicentre multi-device hybrid imaging study of coronary artery disease: results from the EValuation of INtegrated Cardiac Imaging for the Detection and Characterization of Ischaemic Heart Disease (EVINCI) hybrid imaging population. Eur Heart J Cardiovasc Imaging. 2016 Sep;17(9):951-60. doi: 10.1093/ehjci/jew038. Epub 2016 Mar 18. PMID 26992419
- [Background] Mutuberria-Urdaniz M, Pizzi MN, Aguade-Bruix S, Candell-Riera J, Otaegui-Irurueta I. [Spastic coronary artery. Correlation of the myocardium at risk with scintigraphy and coronary angiography]. Rev Esp Med Nucl Imagen Mol. 2013 Jan;32(1):40-2. doi: 10.1016/j.remn.2011.12.004. Epub 2012 May 8. Spanish. PMID 23177343
- [Background] Weber KT. What can we learn from exercise testing beyond the detection of myocardial ischemia? Clin Cardiol. 1997 Aug;20(8):684-96. doi: 10.1002/clc.4960200805. PMID 9259161
- [Background] Candell-Riera J, Santana-Boado C, Castell-Conesa J, Aguade-Bruix S, Bermejo-Fraile B, Soler-Soler J. Dipyridamole administration at the end of an insufficient exercise Tc-99m MIBI SPECT improves detection of multivessel coronary artery disease in patients with previous myocardial infarction. Am J Cardiol. 2000 Mar 1;85(5):532-5. doi: 10.1016/s0002-9149(99)00806-1. PMID 11078262
- [Background] Candell-Riera J, Santana-Boado C, Castell-Conesa J, Aguade-Bruix S, Olona M, Palet J, Cortadellas J, Garcia-Burillo A, Soler-Soler J. Simultaneous dipyridamole/maximal subjective exercise with 99mTc-MIBI SPECT: improved diagnostic yield in coronary artery disease. J Am Coll Cardiol. 1997 Mar 1;29(3):531-6. doi: 10.1016/s0735-1097(96)00562-1. PMID 9060889
- [Background] Johnson SG, Peters S. Advances in pharmacologic stress agents: focus on regadenoson. J Nucl Med Technol. 2010 Sep;38(3):163-71. doi: 10.2967/jnmt.109.065581. Epub 2010 Aug 19. PMID 20724531
- [Background] Cassar A, Chareonthaitawee P, Rihal CS, Prasad A, Lennon RJ, Lerman LO, Lerman A. Lack of correlation between noninvasive stress tests and invasive coronary vasomotor dysfunction in patients with nonobstructive coronary artery disease. Circ Cardiovasc Interv. 2009 Jun;2(3):237-44. doi: 10.1161/CIRCINTERVENTIONS.108.841056. Epub 2009 May 8. PMID 20031721
- [Background] Rodriguez-Sinovas A, Sanchez JA, Gonzalez-Loyola A, Barba I, Morente M, Aguilar R, Agullo E, Miro-Casas E, Esquerda N, Ruiz-Meana M, Garcia-Dorado D. Effects of substitution of Cx43 by Cx32 on myocardial energy metabolism, tolerance to ischaemia and preconditioning protection. J Physiol. 2010 Apr 1;588(Pt 7):1139-51. doi: 10.1113/jphysiol.2009.186577. Epub 2010 Feb 15. PMID 20156849
- [Background] Caselli C, Rovai D, Lorenzoni V, Carpeggiani C, Teresinska A, Aguade S, Todiere G, Gimelli A, Schroeder S, Casolo G, Poddighe R, Pugliese F, Le Guludec D, Valente S, Sambuceti G, Perrone-Filardi P, Del Ry S, Marinelli M, Nekolla S, Pietila M, Lombardi M, Sicari R, Scholte A, Zamorano J, Kaufmann PA, Underwood SR, Knuuti J, Giannessi D, Neglia D; EVINCI Study Investigators. A New Integrated Clinical-Biohumoral Model to Predict Functionally Significant Coronary Artery Disease in Patients With Chronic Chest Pain. Can J Cardiol. 2015 Jun;31(6):709-16. doi: 10.1016/j.cjca.2015.01.035. Epub 2015 Feb 2. PMID 26022987
- [Background] Barba I, Jaimez-Auguets E, Rodriguez-Sinovas A, Garcia-Dorado D. 1H NMR-based metabolomic identification of at-risk areas after myocardial infarction in swine. MAGMA. 2007 Dec;20(5-6):265-71. doi: 10.1007/s10334-007-0097-8. Epub 2007 Dec 20. PMID 18095012
- [Background] Barba I, de Leon G, Martin E, Cuevas A, Aguade S, Candell-Riera J, Barrabes JA, Garcia-Dorado D. Nuclear magnetic resonance-based metabolomics predicts exercise-induced ischemia in patients with suspected coronary artery disease. Magn Reson Med. 2008 Jul;60(1):27-32. doi: 10.1002/mrm.21632. PMID 18581408